CLINICAL TRIAL: NCT01611350
Title: Behavior Change Interventions to Improve the Acquisition and Correct Use of Improved Cookstoves
Brief Title: Testing New Marketing Models for Improved Cookstoves - Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Impact Carbon, 501c3 (Unknown); Centre for Integrated Research and Community Development Uganda (CIRCODU) (Unknown)
Responsible Party: Principal Investigator, Theresa Beltramo, Principal Investigator, University of California, Berkeley
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TRA001
Record Dates: First submitted 2012-02-08; First posted 2012-06-05 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Air Pollution, Indoor; Behavior
Keywords: Indoor Air Pollution; Marketing Methods for Increasing Technology Adoption; Optimal Contracts for Technology Adoption
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: We conducted a series of sequential RCTs. The first RCT tests how willingness to pay for a fuel-efficient cookstove varies with 1. marketing messages and 2. sales offers that address household financial constraints The second RCT 2 tests the comparable purchase from a traditional cash-and carry sales offer to uptake of the novel offer- which includes a free trial of the cookstove and the right to return the stove with no payment and a rent-to-own model where the customer pays in time payments.
  The third RCT examined the effects of fuel-efficient cookstoves on wood use, household air pollution, and cooking behaviors in rural Uganda RCT 4 examines the effect of peer usage on consumer demand for efficient cookstoves with a randomized controlled trial in rural Uganda.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Health Marketing Message (Experimental): Marketing message focused on health effects of cooking with wood on a three stone fire.
  Interventions: Other: RCT 1- Testing the Effectiveness of Marketing Messages in Increasing Willingness to Pay
- Savings Marketing Message (Experimental): Marketing message focused on savings (both time and money) related to using an energy efficient cookstove.
  Interventions: Other: RCT 1- Testing the Effectiveness of Marketing Messages in Increasing Willingness to Pay
- Savings and Health Marketing Messages Combined (Experimental): One group will receive both the savings and health marketing messages.
  Interventions: Other: RCT 1- Testing the Effectiveness of Marketing Messages in Increasing Willingness to Pay
- Novel Sales Offer (Experimental): This group will receive a free trial and time payments when purchasing an energy efficient cookstove.
  Interventions: Other: RCT 2- Testing the Effectiveness of the Novel Sales Offer and its ability to Increase Uptake of Purchasing Energy Efficient Cookstoves
- Early vs. Late Buyers (Experimental): Of those who accept the Novel Sales Offer, half the buyers will randomly be selected to start their free trial within a few weeks of the sales meeting, while the other half- the late buyers- will start their free trial a within 2 months of the sales meeting.
  Interventions: Other: RCT 3-Measure the Effects of Fuel Efficient Cookstoves on Health, Fuel Use and Time Spent Collecting Fuel

INTERVENTIONS:
Other: RCT 1- Testing the Effectiveness of Marketing Messages in Increasing Willingness to Pay — We are testing whether any marketing messages effect participants willingness to pay for the fuel efficient cookstoves. All marketing messages are true.
  Arms: Health Marketing Message; Savings Marketing Message; Savings and Health Marketing Messages Combined
Other: RCT 3-Measure the Effects of Fuel Efficient Cookstoves on Health, Fuel Use and Time Spent Collecting Fuel — Of those who accept the Novel Sales Offer, half the group will be randomly selected to start their free trial early while the other half will receive their free trial late. Those who receive their free trial late will serve as a control group for fuel consumption and Particulate Matter exposure in kitchens.
  Arms: Early vs. Late Buyers
Other: RCT 2- Testing the Effectiveness of the Novel Sales Offer and its ability to Increase Uptake of Purchasing Energy Efficient Cookstoves — We are testing whether households who receive the Novel Sales Offer have higher uptake than those households who receive the Traditional Sales Offer.
  Arms: Novel Sales Offer

SUMMARY:
The purpose of this study is to determine the effectiveness of different sales offers and different marketing messages to increase the uptake of energy efficient cookstoves.

This research will address the following major barriers to the acquisition and correct use of improved cookstoves into four main categories:

* Inappropriate product or marketing for intended users
* Lack of consumer trust in new products
* Failure to address consumers' financial constraints
* Failure to achieve behavioral change

To do so this research includes 3 Randomized Controlled Trials including:RCT 1- Testing the Effectiveness of Marketing Messages in Increasing Willingness to Pay; RCT 2- Testing the Effectiveness of the Novel Sales Offer and its ability to Increase Uptake of Purchasing Energy Efficient Cookstoves; and RCT 3-Measure the Effects of Fuel Efficient Cookstoves on Health, Fuel Use and Time Spent Collecting Fuel.

RCT 1 studies the price women are willing to pay for the improved stove. It will also test the effects of the two most effective marketing messages identified during the Phase 1 Feasibility stage (e.g., improved health, saves time, and has high status) on increasing willingness to pay. RCT 1 will run second price auctions in 36 parishes with an average of 60 participants per meeting.

From RCT 1, RCT 2 tests the effect of a Novel Sales Offer- which includes a free trial, and time payments- on purchasing decisions of participants versus those that receive the Traditional Offer- a cash and carry offer. Based on a pilot in urban Kampala conducted by Dr. David I. Levine (co-P.I. on this project) results show a 44% uptake for households offered the novel offer vs. a 4% uptake for those offered the traditional offer. The hypothesis is a novel offer will significantly increase uptake of fuel efficient cookstoves in rural Uganda when compared to a traditional offer.

RCT 3 measures the impacts of fuel efficient cookstoves on health, fuel usage, and time spent collecting fuel. For RCT 3 we will randomize those who accept the Novel Offer into early and late groups. To measure the impacts of improved stoves on health, fuel use, time spent collecting fuel, etc., there will be a baseline and follow-up survey and associated quantitative measures on our full sample and a small endline on select quantitative measures for a sub-sample.

DETAILED DESCRIPTION:
Given that 95% of Ugandans rely on solid fuel for cooking, and the vast majority use unimproved wood stoves in rural areas, replacing dirty and inefficient household wood stoves in Uganda provides a tremendous opportunity to improve health. Impact Carbon has been implementing an improved cookstove program in Uganda since 2005 which has now commercially sold more than 80,000 stoves. However, the program has not been successful in selling clean burning household wood stoves due to challenges related to the four categories of major barriers discussed above. Targeted research addressing these barriers will allow the team to test new sales and marketing methods to increase uptake of fuel efficient cookstoves. This has the potential to significantly reduce indoor air pollution as more households adopt fuel efficient cookstoves.

ELIGIBILITY:
All households are eligible to purchase a stove.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2012-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Marketing Messages in Increasing Willingness to Pay | During February 2012 we will assess whether or not different marketing messages increase willingness to pay.
  We will test whether or not certain marketing messages increase willingness to pay through a secondary price auction.

SECONDARY OUTCOMES:
Test the Effectiveness of the Novel Sales Offer to Increase Uptake of Purchasing Energy Efficient Cookstoves | This will be assessed from March 2012 to July 2012
  We will randomly select some parishes to receive the Novel Sales Offer which includes a free trial and time payments and some parishes to receive the Traditional Offer, which is the offer to pay full price immediately. The outcome will be the percentage of both groups which accept the Novel Offer vs. those that accept the Traditional Offer.
Measure the Effects of Fuel Efficient Cookstoves on Health, Fuel Use and Time Spent Collecting Fuel | Will be assessed between April 2012 and August 2012
  We will measure wood use by weighing wood before without fuel efficient stove and after with fuel efficient stove.
  To monitor effects on health we will measure Particulate Matter via. UCB PATS monitors. We will measure PM before without the fuel efficient stove and after with the fuel efficient stove.
  We will measure time spent collecting fuel by self reporting survey questions from a baseline, follow-up and endline survey.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Beltramo, PhD, Principal Investigator — University of California, Berkeley
Locations (2):
- Haas School of Business, University of California, Berkeley, Berkeley, California, United States
- Mbarara District, Mbarara, Uganda

REFERENCES:
- See also: Published article for RCT 1: "The effect of marketing messages and payment over time on willingness to pay for fuel-efficient cookstoves — https://ideas.repec.org/a/eee/jeborg/v118y2015icp333-345.html